CLINICAL TRIAL: NCT06667284
Title: Gastroduodenal Intussusception: Two Cases of Gastroduodenal Intussusception Following Gastric Plication, Each Managed with a Different Approach.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ibn Al Nafees Hospital (Other Government)
Collaborators: Damascus University (Other)
Responsible Party: Principal Investigator, Yamen Madi, General surgeon, Damascus University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Gastroduodenal intussuception
Record Dates: First submitted 2024-10-28; First posted 2024-10-31 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-10

CONDITIONS: Bariatric Surgery; Intussusception
Keywords: case report; gastric plication
MeSH Terms: conditions — Intussusception

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group a (Active Comparator): Roux en y procedure
  Interventions: Procedure: Roux en y procedure
- Group b (Active Comparator): Omega Brown anastomosis
  Interventions: Procedure: Omega brown procedure

INTERVENTIONS:
Procedure: Roux en y procedure — subtotal gastrectomy en bloc with Roux-en-Y reconstruction, using TA 90 and GIA staplers. The length of the biliopancreatic limb was 50 cm, while the alimentary limb was 80 cm
  Arms: Group a
Procedure: Omega brown procedure — Gastrojejunal anastomosis with jejunojejunal anastomosis
  Arms: Group b

SUMMARY:
The investigators received two female patients in the hospital who developed gastroduodenal intussusception following gastric plication procedure, requiring surgical treatment. Both patients presented with non-specific, atypical abdominal pain several months after the gastric plication. Both patients required surgical intervention, which included manual reduction of the plication followed by subtotal gastrectomy en bloc with Roux-en-Y reconstruction. In the second case, an Omega Brown anastomosis was performed, and a jejunostomy was created after the anastomosis in both patients.

ELIGIBILITY:
Inclusion Criteria:

- Patients with gastro-duodenal intussusception following a gastric plication procedure.

Exclusion Criteria:

* children

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Estimated)
Dates: Start 2024-10-31 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-01-15 (Estimated)

PRIMARY OUTCOMES:
Comparison of management strategies for gastro-duodenal intussusception following gastric plication. | 12 weeks following end of treatment.
  The investigators compare the outcomes of managing bowel obstruction and abdominal pain after each surgery. The Investigator use small bowel obstruction prediction score index

REFERENCES:
- [Background] Coco D, Leanza S, Fiume I. Small bowel obstruction: a prognostic score index for surgery - a review. Prz Gastroenterol. 2022;17(3):177-182. doi: 10.5114/pg.2022.118454. Epub 2022 Aug 3. PMID 36127935